CLINICAL TRIAL: NCT00648687
Title: Evaluation of the Pain Response During Examination for Retinopathy of Prematurity in Very Low Birth Weight Infants
Brief Title: Pain Response During Examination for Retinopathy of Prematurity
Acronym: ROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bioethics Commission of Brazil (Other)
Responsible Party: Renato Procianoy, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HCPA 07437
Record Dates: First submitted 2008-03-14; First posted 2008-04-01 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-09

CONDITIONS: Retinopathy of Prematurity
Keywords: prematurity; retinopathy of prematurity; pain; very low birth weight infants
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth; Pain | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): this group will receive oral water and glucose prior to eye exam
  Interventions: Behavioral: suck 12.5% dextrose in water 5 minutes before the procedure
- II (No Intervention): this group is the control group.

INTERVENTIONS:
Behavioral: suck 12.5% dextrose in water 5 minutes before the procedure — Newborns will suck 2 ml of D12.5W 5 minutes before eye exam for ROP
  Arms: I

SUMMARY:
Newborns infants equal or less than 1500 grams and/or equal and less than 32 weeks will have ophthalmologic examination for ROP at 6 weeks old. They will be randomized blindly to receive 2 ml of 12.5% dextrose in water (D12.5W) orally five minute before examination (intervention group) or nothing (control). NIPS scale will be applied two minutes before examination and two minutes after examination.

ELIGIBILITY:
Inclusion Criteria:

* all newborns equal or less than 1500 grams birth weight and/or equal or less than 32 weeks gestational age

Exclusion Criteria:

* the ones that died before 6 weeks old

Ages: 5 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pain secondary to eye examination | 2 minutes after the exam

CONTACTS AND LOCATIONS:
Overall Officials: Renato S Procianoy, MD,PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Costa MC, Eckert GU, Fortes BG, Fortes Filho JB, Silveira RC, Procianoy RS. Oral glucose for pain relief during examination for retinopathy of prematurity: a masked randomized clinical trial. Clinics (Sao Paulo). 2013;68(2):199-204. doi: 10.6061/clinics/2013(02)oa13. PMID 23525316